CLINICAL TRIAL: NCT01570491
Title: Cardiothoracic Anesthesia and Critical Care Patient Registry
Brief Title: A Real-Time Ultrasound Guided Approach For Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-1171
Record Dates: First submitted 2012-03-27; First posted 2012-04-04 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Patients Aged 55 or Older; BMI More Than 40 kg/m2; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound-guided spinal anesthesia (Active Comparator): participants will randomly assigned to use ultrasound-guided technique for block placement by Anesthesiologist.
  Interventions: Other: ultrasound-guided spinal anesthesia
- standard spinal anesthesia (Placebo Comparator): randomized participants will be given standard spinal anesthesia insertion technique for block placement by Anesthesiologist
  Interventions: Other: standard spinal anesthesia

INTERVENTIONS:
Other: ultrasound-guided spinal anesthesia — ultrasound-guided technique for block placement
  Arms: ultrasound-guided spinal anesthesia
Other: standard spinal anesthesia — Anesthesiologist will use standard technique for placement of spinal block.
  Arms: standard spinal anesthesia

SUMMARY:
Our goal was to compare the number of attempts to perform spinal anesthesia using real-time ultrasound guidance versus landmark technique in patients meeting predefined criteria for difficult spinal anesthesia.

DETAILED DESCRIPTION:
Patients who consent to receive spinal anesthesia (as opposed to some other anesthetic technique) and who meet the inclusion/exclusion criteria for the study (given below) will be randomized on day of surgery after obtaining informed consent to either ultrasound-guided or standard spinal anesthesia technique.

A block randomization scheme with random block sizes ranging from 2-8 patients will be used. The outcomes will be recorded by a third party observer in the block room/operating room who might be a nurse or resident or clinical research fellow not directly involved with performing the block. The post procedure outcomes will also be recorded by a clinical research fellow or resident who was not directly involved with performing the block.

No sample size estimation methodology currently exists for the right-censored count data models. We expect less number of attempts in the ultrasound group a 20 % difference between the two groups which we feel is a minimum of a clinically-relevant effect. At the 0.05 level of significance with a power of 0.8, we will require a minimum of 20 patients per group,therefore we plan to recruit 40 patients in total.

The analysis will be conducted by a statistician who will be blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 55 or older
2. BMI more than 40
3. Scoliosis

Exclusion criterion:

1 Patients who have undergone previous Spine Surgery

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Elsharkawy, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were recruited and enrolled from 4/2012 to 10/2012 at Cleveland clinic, main campus.
Groups:
- Ultrasound-guided Spinal Anesthesia: Anesthesiologist will use ultrasound-guided technique for spinal anesthesia block placement.
  ultrasound guided placement spinal block: Anesthesiologist will use ultrasound as a guide for placement of spinal block.
- Standard Spinal Anesthesia: Anesthesiologist will use standard spinal anesthesia insertion technique for block placement.
  standard spinal anesthesia: Anesthesiologist will use standard technique for placement of spinal block.
Period: Overall Study
Arm/Group | Ultrasound-guided Spinal Anesthesia | Standard Spinal Anesthesia
Started | 19 | 19
Completed | 14 | 18
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — treatment: not given or discontinued | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound-guided Spinal Anesthesia | Standard Spinal Anesthesia | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10) | 70 (10) | 70 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Attempts
Description: Number of attempts (defined as number of needle reinsertions form the skin and NOT number of redirection of the needle) at the beginning of surgery
Time Frame: 10-15 minutes before the surgery
Measure: Median (Inter-Quartile Range); unit: Attempts
Arm/Group | Ultrasound-guided Spinal Anesthesia | Standard Spinal Anesthesia
Number analyzed (Participants) | 14 | 18
Attempts | 1 [1 to 2] | 1 [1 to 2]
Statistical Analysis 1: Comparison: Ultrasound-guided Spinal Anesthesia vs Standard Spinal Anesthesia; We hypothesized that real-time US guidance would result in a 20% lower number of attempts compared to the control group. At the 0.05 level of significance with a power of 0.8, we will require a minimum of 20 patients per group, therefore we planned to recruit 40 patients in total; Test type: Superiority or Other; p = 0.83, Kruskal-Wallis

2. Secondary Outcome: Difficulty of Block Insertion
Description: Difficulty of insertion, was rated by the performing anesthesiologist on a 10-point Likert scale from one (easy) to ten (extremely difficult)
Time Frame: 10-15 minutes before the surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ultrasound-guided Spinal Anesthesia | Standard Spinal Anesthesia
Number analyzed (Participants) | 14 | 18
units on a scale | 5.5 [4 to 7] | 2.5 [2 to 4]
Statistical Analysis 1: Comparison: Ultrasound-guided Spinal Anesthesia vs Standard Spinal Anesthesia; Test type: Superiority; p = 0.001, Kruskal-Wallis

3. Secondary Outcome: Patient Satisfaction
Description: Record patient satisfaction on a five-point Likert scale, where a value of 1 indicates extremely unsatisfied and a value of 5 indicates extremely satisfied.
Time Frame: after insert the block but before the surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ultrasound-guided Spinal Anesthesia | Standard Spinal Anesthesia
Number analyzed (Participants) | 14 | 18
units on a scale | 5 [4 to 5] | 5 [5 to 5]
Statistical Analysis 1: Comparison: Ultrasound-guided Spinal Anesthesia vs Standard Spinal Anesthesia; Test type: Superiority; p = 0.09, Kruskal-Wallis

4. Secondary Outcome: Time to Perform Block (Second)
Description: Time to perform block (from first needle insertion to injection of medication)
Time Frame: as measured in seconds after needle insertion, surgical date
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Ultrasound-guided Spinal Anesthesia | Standard Spinal Anesthesia
Number analyzed (Participants) | 14 | 18
second | 117.5 [67 to 247] | 256 [144 to 327]
Statistical Analysis 1: Comparison: Ultrasound-guided Spinal Anesthesia vs Standard Spinal Anesthesia; Test type: Superiority; p = 0.06, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: from date of surgery to hospital discharge, on average of 1 week
Arm/Group | Ultrasound-guided Spinal Anesthesia | Standard Spinal Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 0/14 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No